CLINICAL TRIAL: NCT00348010
Title: Double-blind, Randomized, Dose-titration, Parallel-group Comparison of the Efficacy and Safety of Extended Release Tramadol Hydrochloride (Tramadol HCl ER) and Placebo in the Treatment of Osteoarthritis of the Knee.
Brief Title: A Study Comparing the Effectiveness and Safety of Extended Release Tramadol Versus Placebo for the Treatment of Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B00.CT3.015.TRA PO3
Record Dates: First submitted 2006-07-02; First posted 2006-07-04 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Pain
Keywords: osteoarthritis; knee pain; extended release analgesia; opioid
MeSH Terms: conditions — Chronic Pain; Osteoarthritis

INTERVENTIONS:
Drug: Tramadol HCl ER

SUMMARY:
The purpose of this study is to compare the analgesic effectiveness and safety of tramadol HCl ER to placebo in patients with moderate to severe pain due to osteoarthritis (OA). The study hypothesis is that tramadol HCl ER is effective and safe in the treatment of OA.

DETAILED DESCRIPTION:
Immediate release (IR) tramadol has demonstrated efficacy in several pain conditions including: obstetrical, gynecological, orthopedic, abdominal, and oral surgery. The short elimination half-life of IR tramadol requires every 4-6 hour dosing to maintain optimal levels of analgesia in chronic pain. The study medication in this study is a once-daily, extended-release (ER) tramadol formulation. This is a 12-week, multi-center, double-blind, randomized, dose-titration, parallel-group, placebo-controlled study designed to evaluate the analgesic effectiveness and safety of once daily tramadol HCl ER with placebo in the treatment of patients with OA of the knee. Patients with OA Functional Class I-III of the knee will be eligible for participation, if appropriate criteria are met. After a 2-7 day washout period, during which the use of all analgesic medications used for chronic pain management will be discontinued, patients experiencing moderate to severe pain (pain intensity >= 40 mm on a 100 mm visual analog scale) in the index knee and who meet all other study criteria will enter a 2-week, double-blind, titration period. During this period, patients will be randomly assigned to treatment with tramadol HCl ER or placebo, once daily (QD). The initial dose will be tramadol HCl ER 100 mg or matching placebo QD. On Day 4 and for the remainder of the week, patients will be titrated to 200 mg or matching placebo QD, based on tolerability. Beginning at Visit 3, a minimum dose of 200 mg or matching placebo QD are to be maintained for the remainder of the 12-week study. Patients unable to tolerate at least 200 mg or matching placebo QD will be discontinued from the study. After Week 1 (Visit 3), further increases to 300 mg or 400 mg or matching placebo QD were permitted, depending on the adequacy of pain relief and tolerability of side effects. Efficacy and safety evaluations will be collected at study visits occurring at Weeks 1, 2, 4, 8, and 12 or at early termination. Study medication will be discontinued at Week 12 and patients will return after 1 week for a post-treatment visit (Week 13).

ELIGIBILITY:
Inclusion Criteria:

* Patients with American College of Rheumatology (ACR) Functional Class I-III OA of the knee; involvement of at least one knee joint that warrants treatment with NSAIDs, acetaminophen, or opioid analgesics for at least 75 of the 90 days preceding the screening visit; patients with radiographic evidence of osteoarthritis within the last 6 months; patients with a pain intensity in index joint > = 40 mm on the visual analog scale (VAS) at the baseline visit; patients who are able to discontinue NSAIDs, COX-2 selective inhibitors, and other analgesics during the washout period and throughout double-blind study.

Exclusion Criteria:

* Patients with a medical condition, other than OA, uncontrolled with treatment or any clinically significant condition that, in the investigator's opinion, precludes study participation or interferes with the assessment of chronic pain and other OA symptoms; patients with a diagnosis of inflammatory arthritis, gout, pseudo-gout or Paget's disease, that, in the investigator's opinion, interferes with the assessment of pain and other symptoms of OA; patients with a diagnosis of chronic pain syndrome, patients with an ACR or a clinical diagnosis of fibromyalgia; patients with a clinically significant form of joint disease or prior joint replacement surgery at the index joint; patients with an anticipated need for surgery or other invasive procedure in the index joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245
Dates: Start 2000-11; Study Completion 2001-07

PRIMARY OUTCOMES:
The primary efficacy outcome is the change in arthritis pain intensity score
averages over the 12 weeks of the study.

SECONDARY OUTCOMES:
The secondary outcomes include change from baseline in the daily arthritis
pain intensity VAS score from patient diaries; WOMAC OA Index pain subscale
scores for pain and physical function, patient's global assessment, patient's
sleep assessment

REFERENCES:
- [Background] Babul N, Noveck R, Chipman H, Roth SH, Gana T, Albert K. Efficacy and safety of extended-release, once-daily tramadol in chronic pain: a randomized 12-week clinical trial in osteoarthritis of the knee. J Pain Symptom Manage. 2004 Jul;28(1):59-71. doi: 10.1016/j.jpainsymman.2003.11.006. PMID 15223085